CLINICAL TRIAL: NCT03612401
Title: Treatment of Spinal Cord Injury Patients for Neurogenic Bladder: an Open Label Pilot Study of Anticholinergic Agent vs. Mirabegron (MYRBETRIQ ®) to Evaluate Cognitive Impact and Efficacy
Brief Title: Treatment of Spinal Cord Injury Patients for Neurogenic Bladder: Anticholinergic Agent vs. Mirabegron
Acronym: SCIMYR
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20180376H
Record Dates: First submitted 2018-07-09; First posted 2018-08-02 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Spinal Cord Injuries; Neurogenic Bladder; Cognitive Change
Keywords: Spinal cord injury; SCI; Neurogenic bladder; Overactive bladder; anticholinergic; mirabegron; cognitive; cognition; NGB; OAB
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic; Urinary Bladder, Overactive | interventions — mirabegron

STUDY DESIGN:
Intervention Model Description: Open label, pilot study comparing baseline measurement anticholinergic agent vs. study intervention mirabegron (MYRBETRIC ®) to evaluate cognitive impact and efficacy (SCIMYR)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neurogenic Bladder (Other): Spinal Cord Injury patients with known neurogenic bladder on treatment with Anticholinergic Agents at baseline switched to mirabegron as the study intervention
  Interventions: Drug: Mirabegron

INTERVENTIONS:
Drug: Mirabegron — Beta-3 adenoreceptor agonist
  Other Names: MYRBETRIQ

SUMMARY:
We propose to test the hypothesis that cognition will improve with substitution of mirabegron for the anticholinergic agent (AC) in elderly persons with spinal cord injury (SCI) who require neurogenic bladder (NGB) treatment.

DETAILED DESCRIPTION:
The strong evidence for detrimental effects of AC agents on cognition, led the American Urological Association to update its guidelines in 2015 to include mirabegron as an alternative first-line agent for treatment of overactive bladder (OAB). NGB symptoms are very similar to OAB so the conditions are often treated similarly; however, data is lacking on the use of this promising agent for NGB. We thus propose to test the hypothesis that cognition will improve with substitution of mirabegron for the AC agent in elderly persons with SCI who require NGB treatment.

Subjects eligible for enrollment will have been treated with an anticholinergic agent for at least 3 months prior to enrollment. Baseline measurements will be recorded for subjects currently treated with an AC agent, after enrollment, the subject will start treatment with the study drug. Measurements from baseline (AC agent) will be compared to measurements taken after study intervention (mirabegron).

ELIGIBILITY:
Inclusion Criteria:

1. Both genders with spinal cord injury being treated for neurogenic bladder and age >60 years
2. All ethnic groups
3. Veterans will be enrolled to allow mailing of study medication by VA pharmacies.
4. Laboratory results:

   Normal clinical labs for CBC (complete blood count), CMP (comprehensive metabolic panel), and UA (urinalysis) within past 6 months or repeat at screening if none. For example: HCT (hematocrit) ≥34%, GFR (glomerular filtration rate) ≥ 30 mL/min, liver enzymes (AST (aspartate aminotransferase test) < 2 x upper limit of normal, ALT (alanine aminotransferase test) < 2 x upper limit of normal, alkaline phosphatase < 2 X upper limit of normal), normal electrolytes, urinalysis and asymptomatic for UTI (urinary tract infection)
5. Taking a minimum regimen for 3 months of anticholinergic agent.

Exclusion Criteria:

1. Diagnosis of dementia or cognitive impairment from another condition such as TBI (traumatic brain injury), ALZ (alzheimers), Lewy body dementia or vascular dementia
2. End stage renal disease (GFR <30) or bladder obstruction
3. Poorly controlled blood pressure (BP), systolic BP>180, diastolic BP>110 mmHg)
4. Renal function - exclude if serum creatinine >2x normal range
5. Liver function - exclude if >2x normal liver enzyme levels
6. History of, or currently active treatment for cardiac dysrhythmias, including atrial fibrillation (eg. apixaban. If subject is currently taking metoprolol they will be monitored and dose may need to be adjusted on mirabegron)
7. Current treatment with desipramine, digoxin
8. Active/unstable conditions: inflammatory, thyroid, autoimmune, gastrointestinal (GI), hematologic, or neoplastic disorders. Exclude subjects with clinical lab values outside the normal range (other than as specified above).
9. Subject is considered unsuitable for the study in the opinion of the investigator for any other reason

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in cognitive measure - Logical Memory I (Immediate) - baseline and post treatment with mirabegron | Change from Week 0 to Week 26
  Wechsler Memory Scale, 4th edition (WMS-IV) subtest

SECONDARY OUTCOMES:
Change in cognitive measure of memory (SLUMS) - baseline and post treatment with mirabegron | Change from Week 0 to Week 26
  Saint Louis University Mental Status Exam (SLUMS) - a series of shapes and recall measures
Change in cognitive measure of executive function (Stroop test) - baseline and post treatment with mirabegron | Change from Week 0 to Week 26
  Stroop Color and Word Test - a series of color-word and picture-word tests of executive function
Change in cognitive measure of executive function (SDMT) - baseline and post treatment with mirabegron | Change from Week 0 to Week 26
  Symbol Digit Modalities Test - a series of symbols to assess executive function
Change in memory and executive function (TEXAS) - baseline and post treatment with mirabegron | Change from Week 0 to Week 26
  Texas Executive Assessment (TEXAS) - A series of short term recall measures
Change in Neurogenic Bladder Symptom Score (NBSS) - baseline and post treatment with mirabegron | Change from Week 0 to Week 26
  Neurogenic bladder symptom questionnaire
Change in Neurogenic Bowel Dysfunction Score (NBD) - baseline and post treatment with mirabegron | Change from Week 0 to Week 26
  Neurogenic bowel questionnaire
Change in cognitive measure - Logical Memory II (Delayed) - baseline and post treatment with mirabegron | Change from Week 0 to Week 26
  Wechsler Memory Scale, 4th edition (WMS-IV) subtest

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Trbovich, MD, Principal Investigator — UT Health San Antonio and VA Spinal Cord Clinic
Locations (1):
- South Texas Veterans Health Care System, Audie L. Murphy Hospital, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Publication of study results in Spinal cord series and cases. — https://pubmed.ncbi.nlm.nih.gov/34112758/